CLINICAL TRIAL: NCT03850756
Title: New Diagnostic System for the Early Detection of Chronic Renal Damage Associated to Tobacco Consumption: Preventive and Personalized Application
Brief Title: Early Diagnosis of Kidney Damage Associated With Tobacco Use
Status: Completed | Type: Observational
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Grupo de Investigación de Atención Primaria de Castilla y León (Other Government); Salamanca University Hospital (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: BIOTAB
Record Dates: First submitted 2018-12-27; First posted 2019-02-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Kidney Injury; Kidney Disease, Chronic; Tobacco Toxicity
Keywords: Biomarker; Tobacco; Nephrotoxicity; Prevention; Diagnosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In this project, only urine samples will be collected. This will be centrifuged, aliquoted and stored at -80 degrees Celsius until its determination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: No smokers without risk factors: A smoker is defined as: any person who habitually consumes tobacco at the time of taking the sample or who has left it in the last 12 months (WHO, 2008).
  The following circumstances involved in the development of kidney damage will be considered a risk factor: Diabetes Mellitus, Hypertension and / or frequent use of NSAIDs (more than three days a week during the three months prior to sampling)
  In these patients kidney function will be evaluated by:
  Early kidney damage biomarkers Predisposition to kidney injury biomarkers
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Predisposition to kidney injury biomarkers
- 2: No smokers with risk factors: A smoker is defined as: any person who habitually consumes tobacco at the time of taking the sample or who has left it in the last 12 months (WHO, 2008).
  The following circumstances involved in the development of kidney damage will be considered a risk factor: Diabetes Mellitus, Hypertension and / or frequent use of NSAIDs (more than three days a week during the three months prior to sampling)
  In these patients kidney function will be evaluated by:
  Early kidney damage biomarkers
  Interventions: Diagnostic Test: Early kidney damage biomarkers
- 3: Smokers without risk factors: A smoker is defined as: any person who habitually consumes tobacco at the time of taking the sample or who has left it in the last 12 months (WHO, 2008).
  The following circumstances involved in the development of kidney damage will be considered a risk factor: Diabetes Mellitus, Hypertension and / or frequent use of NSAIDs (more than three days a week during the three months prior to sampling)
  In these patients kidney function will be evaluated by:
  Early kidney damage biomarkers Predisposition to kidney injury biomarkers
  Also tobacco consumption will be measured
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Predisposition to kidney injury biomarkers; Diagnostic Test: Tobacco consumption
- 4: Smokers without risk factors: A smoker is defined as: any person who habitually consumes tobacco at the time of taking the sample or who has left it in the last 12 months (WHO, 2008).
  The following circumstances involved in the development of kidney damage will be considered a risk factor: Diabetes Mellitus, Hypertension and / or frequent use of NSAIDs (more than three days a week during the three months prior to sampling)
  In these patients kidney function will be evaluated by:
  Early kidney damage biomarkers
  Also Tobacco consumption will be measured
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Tobacco consumption

INTERVENTIONS:
Diagnostic Test: Early kidney damage biomarkers — In the urine samples of these patients, a series of biomarkers of early kidney damage and / or predisposition to kidney damage will be measured.
  Other Names: albumin; N-acetyl-beta-D-glucosaminidase (NAG); Kidney Injury Molecule-1 (KIM-1); Neutrophil gelatinase-associated lipocalin (NGAL); T-gelsolin
Diagnostic Test: Predisposition to kidney injury biomarkers — In the urine samples of these patients, a series of biomarkers of predisposition to kidney damage will be measured.
  Groups: 1: No smokers without risk factors; 3: Smokers without risk factors
Diagnostic Test: Tobacco consumption — In order to know the degree of tobacco consumption, the biomarker cotinine will be measured in the urine samples of these patients.
  Groups: 3: Smokers without risk factors; 4: Smokers without risk factors

SUMMARY:
Tobacco consumption is associated with the appearance of several pathologies, the best known are Chronic Obstructive Pulmonary Disease, several types of cancer and cardiovascular diseases. However, the association between tobacco and kidney damage is not well defined. Some studies suggest that smoking favors progression to chronic kidney disease (CKD). CKD does not have pharmacological treatment and the only clinical strategies useful so far are dialysis or kidney transplantation. Therefore, knowing if tobacco is involved in this disease is a very relevant fact, since it is a modifiable factor. Of all the risk factors associated with the onset and progression of kidney disease is the only one that can be avoid or eliminated. Therefore quitting smoking could help reduce the incidence of this pathology.

In this project, 3 main objectives were proposed:

1. First: to study the tobacco-CKD association in a more exhaustive way. In a population group (patients who attend a primary care center) the renal function of smokers will be evaluated, comparing it with that of non-smokers with similar characteristics (age, sex, etc). In addition, the presence of certain pathologies that can affect the kidney (diabetes mellitus, hypertension and / or frequent consumption of certain medications) will be taken into account. To evaluate the renal functionality, the markers commonly used in the clinic and other more novel ones will be used (urinary biomarkers of early kidney damage).
2. Second: to assess whether smoking patients will be more likely to suffer kidney damage in the future. This will be done by monitoring the patients mentioned above, for two years. During this time, a group of novel markers (urinary biomarkers of predisposition to kidney damage) that in previous studies have detected susceptibility to kidney damage will be evaluated. It will be determined which one or more of these markers are capable of predicting at time 0 (when the first sample of the patient is taken) the subsequent appearance of renal damage.
3. Third: to study whether stopping smoking reduces the risk of developing CKD. It will be evaluated whether stopping smoking reduces the susceptibility to kidney damage by using the biomarkers mentioned above.

DETAILED DESCRIPTION:
According to the WHO, smoking is the main cause of preventable disease and death, being a known risk factor for the development of cancer, respiratory diseases, cardiovascular diseases, etc. Despite the fact that the first associations between smoking and kidney disease date back to the beginning of the last century, up to the present time, evidence has been scarce and inconclusive in the population without risk factors associated with kidney disease.

The increase in the worldwide prevalence of chronic kidney disease and the notable increase in the incidence of patients reaching the final stage of the same, have alerted health systems and have determined that nephrologists focus more on the identification of potentially modifiable prevention factors. Chronic kidney disease has a very high social and economic cost (almost 10% of the affected population and 3% of total health expenditure), which requires coordinated criteria among health professionals to ensure the best levels of quality in prevention, diagnosis and treatment. In this sense, it is recognized that the key to preventive success is a very early diagnosis that allows intervention when the renal functional reserve has not yet been exhausted and, therefore, the excretory function is not yet compromised. In the clinic, one of the most used tools in the diagnosis of kidney damage is based on the detection in the blood of products of metabolism (creatinine, urea, etc.) that begin to accumulate once the renal excretory capacity begins to decrease. However, when the increase in serum urea and creatinine levels is observed, more than 70% of renal function has been lost. Thus, current trends in diagnosis seek to find sensitive markers, specific, and easy to quantify, that detect incipient pathophysiological events produced in early stages, when the damage is less widespread.

To evaluate in depth the association between tobacco consumption and kidney damage, as well as the capacity to recover renal function after cessation of consumption, a longitudinal prospective observational study is proposed. Participants will be informed of the objectives of the project and its benefits both verbally and in writing and will have to sign an informed consent in accordance with the Declaration of Helsinki and the WHO standards for observational studies. Patients will be included completely anonymously and their data will be treated confidentially according to the current data protection legislation. Patients may withdraw freely from the study at any time.

In this study, three main objectives have been proposed:

OBJECTIVE 1: To detect subclinical renal damage in smokers through a battery of early markers.

Previously it was carried out a pilot study with 200 patients in order to check if certain early biomarkers of kidney damage, were able to evidence a possible early lesion not detectable with the usual techniques. The results showed an association between tobacco and kidney damage that needs to be confirmed with a greater number of patients. Based on these results, a new study is considered more robust in terms of the number of patients and broader in terms of the determined markers. It is estimated to include a total of 500 patients (125 per group). The grouping of the same will be based on whether they smoke or not and also be taken into account if they have certain risk factors associated with the onset of kidney damage. Therefore, they will be divided into four groups: 1-No smokers without risk factors, 2-No smokers with risk factors, 3-Smokers without risk factors, 4-Smokers with risk factors.

At the time of inclusion in the study, each patient will obtain the following information: date of collection of the sample; general data (age, sex, drug consumption); anthropometric measurements (body weight, height, body mass index) and analytical biochemistry (plasma creatinine and urea). Information will also be obtained on risk factors for kidney damage (hypertension, diabetes, cardiovascular disease or chronic pain with frequent use of NSAIDs, including the date of diagnosis, the prescribed drugs); tobacco use, the patient will fill out a questionnaire adapted from the WHO MONICA study, which will allow us to classify them as a smoker, non-smoker or ex-smoker and also know the number of cigarettes / cigars consumed per day.

After the recruitment, a urine sample will also be taken in order to analyze the presence of biomarkers of early kidney damage. In addition, the concentration of cotinine in urine (nicotine metabolite) will be evaluated, which will allow to know indirectly the consumption of tobacco in smokers and the absence of tobacco in non-smokers.

OBJECTIVE 2: To study if certain predisposing markers (albumin, and others in patent phase), already identified in previous studies, are able to detect in patients who smoke those who are predisposed to suffer acute kidney damage.

The second strategy proposed in this project raises a new concept of intervention even earlier, before the damage occurs. It has been developed an innovative concept: predisposition to kidney injury. It means that different drugs and renal toxins (in completely subtoxic doses) are capable of predisposing, or making more sensitive to experimental animals to acute kidney damage. The relevance of this situation is that individuals apparently unaffected by the adverse effects of a treatment, or by exposure to toxic substances (such as tobacco) could be exposed to develop acute kidney damage. Associated with this condition it have been identified urinary markers. Their clinical application will allow, not only to detect this predisposition, but to stratify the patients in a preventive and personalized way according to the individual risk of each patient as a result of apparently innocuous pharmacological treatments, or exposure to chemical substances.

To respond to this second objective, a follow-up of 2 years will be carried out to patients in groups 1 and 3, that is, to non-smokers, and to smokers both without risk factors. In this way, the information provided by the markers of kidney damage may be associated with tobacco consumption and not with other causes. In this case, it is estimated that the total number of participants will be 100 per group since it is possible that a percentage of patients will be lost during the follow-up phase. At 24 months, patients will come back to the clinic and deliver a urine sample. In these samples and in the collections in the previous objective (0 months or baseline) the predisposition markers described above will be evaluated. The levels of biomarkers of predisposition at the beginning of the study will be related to renal function in the medium term, evaluated by biomarkers of early damage. In addition, the usual clinical parameters (plasma creatinine, creatinine clearance, plasma urea and proteinuria) will be taken into account.

OBJECTIVE 3: To study whether smoking cessation reduces subclinical renal damage and / or predisposition to acute renal damage.

With this objective, it is proposed to study whether renal parameters and markers are restored once smoking cessation ceases. Which would mean, not only that they are a useful tool in terms of diagnosis, but also an efficient preventive measure.

For this purpose, patients from the "Smoking Unit of the University Assistance Complex of Salamanca (CAUSA)" will be recruited. Those patients who agree to participate in the study will deliver a urine sample at the time of inclusion (time 0 or baseline) and also during follow-up at 3, 6 and 12 months. In these urine samples the markers mentioned in the two previous objectives will be determined. The data provided by the markers of both early injury and predisposition will be useful to analyze the evolution of renal function after the cessation of tobacco use. With this information it well be checked if smoking cessation reduces subclinical renal damage and / or the risk of acute renal damage.

As in Objective 1, after the inclusion of the patient, the following data will be obtained: date of collection of the sample; general data, anthropometric measurements, analytical biochemistry, information about risk factors for kidney damage, date of the diagnosis, prescribed drugs, questionnaire adapted from the WHO MONICA study. Other parameters will also be obtained, such as the concentration of carbon monoxide in exhaled air (measured with a co-oximeter) and the concentration of cotinine in the blood.

COLLECTION OF SAMPLES AND PROCESSING Each patient will be assigned a code, so its identity will only be known by the treating physician. Urine samples will be identified under the established code. Once collected (both those of the Primary Care Center and those of the Smoking Unit), they will be transferred to the CAUSA Sample Bank, where they will be centrifuged, aliquoted and stored at -80 degrees Celsius until they are determined.

ANALYSIS OF URINE SAMPLES All the analytical determinations of this study will be carried out in the laboratories of the "Tera-gnostics of Renal and Cardiovascular Diseases" group of the Bio-sanitary Institute of Salamanca (IBSAL). These determinations will be as follows: proteinuria as a clinical marker of damage by Bradford colorimetric method; early markers of kidney damage by colorimetric kits, ELISA and Western Blot; predisposition markers (in patent phase) by Western Blot, ELISA; Tobacco use marker (cotinine in urine) by ELISA. All urinary concentrations of markers will be corrected by urinary creatinine (colorimetric kit).

STATISTIC ANALYSIS A significance level of 0.05 will be used. The data analysis will be performed with STATA 10 and Statistical Package for the Social Sciences (SPSS) 20.0. Different contrasts will be applied depending on the association that is to be studied in each case, and the type of variables, such as: normality test (Kolmogorov-Smirnov, Shapiro-Wilk), frequency comparison (χ2), correlation test (Pearson, Spearman), comparison of means for independent data (ANOVA and Kruskal-Wallis) and repeated measures ANOVA and Wilcoxon test for paired data. Finally, to study simultaneously datasets with several variables measured for each individual or parameter collected, a Multivariate Analysis will be used, such as: regression analysis, general linear models, binary logistic regression and correspondence analysis.

LIMITATIONS OF THE STUDY Although the study follows all the recommendations for observational studies considered in the STROBE statement (STrengthening the Reporting of OBservational studies in Epidemiology), there is a possibility that there are factors that have not been considered. On the other hand, the included variables are biomarkers of early kidney damage and predisposition to acute renal damage induced by certain renal toxins. It is possible that there are other markers (unknown), that are not being analyzed, and that can predict the kidney damage associated with smoking.

CONCLUSION In short, this project addresses two issues of high concern in the health field, which are smoking and chronic kidney disease. From its conceptual basis, it raises the possibility of finding a diagnostic tool for the early detection of chronic kidney damage associated with tobacco consumption, with a preventive purpose in terms of the development of the disease and in a personalized way regarding the hypersensitivity of each patient. . Account for it with a consortium of researchers and clinicians consisting of: 1) experts in markers of kidney damage, 2) clinicians specialized in lifestyles and cardiovascular risk, 3) specialists in smoking.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age who agree to participate in the study and do not comply with any of the exclusion criteria

Exclusion Criteria:

* Patients who are terminally ill; presenting previously diagnosed renal failure
* Patients that during the week prior to the sample collection, or at the time of the sample, have been treated with any of the following drugs: aminoglycosides, cephalosporins, tetracyclines, amphotericin B, cisplatin, cyclosporine, foscarnet, acyclovir, cidofovir, radiological contrasts or any other potentially nephrotoxic drug.
* Patients who do not wish to sign the informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be carried out with the general population, specifically patients who attend a Primary Care consultation (Objectives 1 and 2), and people who come to the Smoking Unit to try to stop smoking (Objective 3)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change of urinary albumin | For objectives 1 and 2 (2 years): 0 and 24 months. For the objective 3 (1 year): 0, 3, 6 and 12 months
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary N-Acetyl-β-D-Glucosaminidase (NAG) | For objectives 1 and 2 (2 years): 0 and 24 months. For the objective 3 (1 year): 0, 3, 6 and 12 months
  It is an enzyme whose urinary excretion is elevated in case of kidney damage. It is capable of detecting damage before the classic plasma creatinin and urea markers. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary Kidney Injury Molecule-1 (KIM-1) | For objectives 1 and 2 (2 years): 0 and 24 months. For the objective 3 (1 year): 0, 3, 6 and 12 months
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary Neutrophil gelatinase-associated lipocalin (NGAL) | For objectives 1 and 2 (2 years): 0 and 24 months. For the objective 3 (1 year): 0, 3, 6 and 12 months
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary T-gelsolin. | For objectives 1 and 2 (2 years): 0 and 24 months. For the objective 3 (1 year): 0, 3, 6 and 12 months
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups.This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary biomarkers of predisposition to kidney injury | For objectives 1 and 2 (2 years): 0 and 24 months. For the objective 3 (1 year): 0, 3, 6 and 12 months
  It is a group of markers that are in patent phase so their names can not be mentioned. They are able to detect the susceptibility to kidney damage before administering a nephrotoxic agent. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.

SECONDARY OUTCOMES:
Percentage of patients with Risk factor's | These data will be collected once, at time 0 (moment of inclusion in the study)
  The percentage of participants who suffer each of the following pathologies / conditions (risk factors), in each study group, will be consulted through the clinical history: diabetes mellitus, hypertension, frequent use of NSAIDs.
Body weight | These data will be collected once, at time 0 (moment of inclusion in the study)
  Body weight will be measured to each patient and expressed in kilograms
Height | These data will be collected once, at time 0 (moment of inclusion in the study)
  The height will be measured to each patient and expressed in meters
Body mass index (BMI) | These data will be collected once, at time 0 (moment of inclusion in the study)
  Weight and height will be combined to report BMI in kg/m^2
Age | These data will be collected once, at time 0 (moment of inclusion in the study)
  Through the year of birth, the patient's age will be calculated, which will be expressed in years.
Sex | These data will be collected once, at time 0 (moment of inclusion in the study)
  Patients will be classified according to sex in Male or Female
Concentration of plasma creatinine | These data will be collected once, at time 0 (moment of inclusion in the study)
  From the analytical biochemistry performed on the patient as part of his usual procedure, the plasma creatinine data will be obtained in mg/dL units.
Concentration of plasma urea | These data will be collected once, at time 0 (moment of inclusion in the study)
  From the analytical biochemistry performed on the patient as part of his usual procedure, the plasma urea data will be obtained in mg/dL units.
Quantitative determination of tobacco consumption | For objectives 1 and 2: 0 and 24 months. For the objective 3: 0, 3, 6 and 12 months.
  The urinary excretion of cotinine (tobacco metabolite) in urine will be measured for which a commercial diagnostic kit (ELISA) will be used and expressed as ng/mL. Additionally, if in the biochemical analysis the concentration of cotinine in blood has been determined, this data will be collected and expressed as ng/mL.
Lung capacity | These data will be collected once, at time 0 (moment of inclusion in the study)
  In objective 3, lung capacity will be evaluated with a co-oximeter, and it will be expressed in parts per million (ppm)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Isabel Morales Martín, PhD, Principal Investigator — University of Salamanca
Locations (2):
- Spain (2):
  - Centro de Salud La Alamedilla, Salamanca
  - Unidad de tabaquismo del CAUSA, Salamanca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prieto M, Vicente-Vicente L, Casanova AG, Hernandez-Sanchez MT, Gomez-Marcos MA, Garcia-Ortiz L, Morales AI; members of the Biomarkers of kidney damage and tobacco. Designing new diagnostic systems for the early detection of tobacco-associated chronic renal damage in patients of a primary care centre in Salamanca, Spain: an observational, prospective study protocol. BMJ Open. 2020 Mar 8;10(3):e032918. doi: 10.1136/bmjopen-2019-032918. PMID 32152160
- [Result] Tascon J, Prieto M, Casanova AG, Sanz FJ, Hernandez Mezquita MA, Barrueco Ferrero M, Gomez-Marcos MA, Garcia-Ortiz L, Vicente-Vicente L, Morales AI, On Behalf Of Biotab Team. Early Diagnosis of Kidney Damage Associated with Tobacco Use: Preventive Application. J Pers Med. 2022 Jun 24;12(7):1032. doi: 10.3390/jpm12071032. PMID 35887529

DOCUMENTS (1):
  • Informed Consent Form (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03850756/ICF_000.pdf